CLINICAL TRIAL: NCT02548416
Title: Peroperative Use of Positive End-expiratory Pressure Prevents Formation of Atelectasis as Studied by Computerised Tomography at End of Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Erland Ostberg, M.D., Region Västmanland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dnr 2015/338
Record Dates: First submitted 2015-09-01; First posted 2015-09-14 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2016-11

CONDITIONS: Atelectasis
Keywords: Atelectasis; Positive End-Expiratory Pressure; Oxygenation; Anaesthesia; Computed tomography
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Positive-Pressure Respiration; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEEP group (Active Comparator): Induction and maintenance of anaesthesia in a conventional manner. Peroperative ventilatory settings using positive end-expiratory pressure.
  Interventions: Procedure: Positive end-expiratory pressure
- Control group zero PEEP (Active Comparator): Induction and maintenance of anaesthesia in a conventional manner. Peroperative ventilatory settings using zero end-expiratory pressure.
  Interventions: Procedure: Control group, zero PEEP

INTERVENTIONS:
Procedure: Positive end-expiratory pressure — Induction of anaesthesia is performed in a conventional manner using a target controlled infusion of propofol and remifentanil. Intubation of the trachea is facilitated by rocuronium.
  As soon as correct position of the endotracheal tube is confirmed, controlled ventilation is started with a tidal volume of 7 mL/kg body weight and a respiratory frequency of 10. The fresh gas flow is set to 1 litre/min with an oxygen mixture of 40%, aiming for an inspired oxygen fraction (FiO2) of 30-35%. Positive end-expiratory pressure is set to 6 or 8 cm H20 (8 if BMI>25) in the intervention group.
  Unless the patient´s SpO2 falls below 90%, the FiO2 remains unchanged throughout the procedure.
  Arms: PEEP group
Procedure: Control group, zero PEEP — Induction of anaesthesia is performed in a conventional manner using a target controlled infusion of propofol and remifentanil. Intubation of the trachea is facilitated by rocuronium. As soon as correct position of the endotracheal tube is confirmed, controlled ventilation is started with a tidal volume of 7 mL/kg body weight and a respiratory frequency of 10. The fresh gas flow is set to 1 litre/min with an oxygen mixture of 40%, aiming for an inspired oxygen fraction (FiO2) of 30-35%. Zero PEEP is used.
  Unless the patient´s SpO2 falls below 90%, the FiO2 remains unchanged throughout the procedure.
  Arms: Control group zero PEEP

SUMMARY:
Atelectasis is common during and after general anaesthesia and a number of interventions have been suggested in order to prevent their formation. The use of Positive End Expiratory Pressure (PEEP) during general anaesthesia has in recent years been questioned.

The investigators hypothesize that the use of PEEP as a single intervention improves oxygenation and prevents atelectasis as investigated by computed tomography compared to a control group with zero PEEP.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, American Society of Anesthesiology (ASA) I-II.
* Patients scheduled for non-abdominal day case surgery under general anaesthesia.

Exclusion Criteria:

* ASA class III or higher.
* Body Mass Index (BMI) 30 or higher.
* Arterial oxygen saturation (SpO2) <96% breathing air.
* Chronic Obstructive Pulmonary Disease (COPD).
* Ischaemic heart disease.
* Known or anticipated difficult airway.
* Active smokers and ex-smokers with a history of more than 6 pack years.
* Need for interscalene or supraclavicular plexus block for postoperative pain relief (risk of phrenic nerve paralysis).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Area of atelectasis expressed as centimeter^2 | Within 1-2 hours, just before emergence from anesthesia.The outcome measure (atelectasis) will be investigated at just one point i.e. end of surgery but before emergence from anaesthesia.
  The area of atelectasis in the lungs is assessed by computed tomography (CT) 5-10 mm above the dome of the right diaphragm and expressed in centimeter^2 and as a percentage of the total lung area in the particular scan.
Measurement of aeras with different aeration in the particular CT scan. | Within 1-2 hours, just before emergence from anesthesia.The outcome measure (atelectasis) will be investigated at just one point i.e. end of surgery but before emergence from anaesthesia.
  The areas of different aeration are assessed by computed tomography (CT) 5-10 mm above the dome of the right diaphragm and expressed in centimeter^2 and as a percentage of the total lung area in the particular scan.

SECONDARY OUTCOMES:
Oxygenation, oxygen tension in arterial blood expressed in kilo Pascal (kPa) | Within 1-2 hours, just before emergence from anesthesia. At end of surgery but before emergence from anaesthesia, at the same time as the lungs are investigated by computed tomography.
  Arterial blood gas samples will be drawn and analyzed at the same time as the computed tomography scan will be undertaken.
Oxygenation, oxygen tension in arterial blood expressed in kilo Pascal (kPa) | Within 2 hours perioperatively, 15 minutes after extubation.
  Arterial blood gas samples will be drawn and analyzed 15 minutes after emergence from anesthesia and extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Edmark, Study Director — Region Västmanland
Locations (1):
- Region Västmanland, Köping, Sweden